8/3/2021 9:37 pm

## **Research Consent Form for Biomedical Research**

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates



Protocol Title: A Phase 2 Study of Capmatinib (INC280) IN NSCLC PATIENTS WITH MET EXON 14 ALTERATIONS OR MET AMPLIFICATION WHO HAVE RECEIVED PRIOR MET INHIBITOR

**DF/HCC Principal Research Doctor / Institution:** Rebecca Suk Heist, MD/Massachusetts General Hospital

**DF/HCC Site-Responsible Research Doctors / Institutions:** Daniel Botelho Costa, MD, PhD, MMSc/Beth Israel Deaconess Medical Center

### A. INTRODUCTION

You are invited to take part in a clinical trial, a type of research study, because you have advanced non-small cell lung cancer with a *MET* exon 14 alteration, where you have already received one or more therapies including a MET inhibitor. This research study is studying capmatinib as a possible treatment for this diagnosis.

For purposes of this research, you will be referred to as a "participant."

It is expected that about 20 people will take part in this research study.

Novartis, a pharmaceutical company, is supporting this research study by providing the study drug and additional funding.

This research consent form explains why this research study is being done, what is involved in participating in the research study, the possible risks and benefits of participation, alternatives to participation, and your rights as a research participant. The decision to participate is yours. If you decide to participate, please sign and date at the end of this form. We will give you a copy so that you can refer to it while you are involved in this research study. If you choose not to participate in this research study, the research doctors will discuss other treatment options with you and/or refer you back to your primary doctor.

We encourage you to take some time to think this over, to discuss it with other people and your primary doctor, and to ask questions now and at any time in the future.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | NCT02750215 | |

| 8/3/2021 9:37 pm | | |
|---------------------------------------|----------------|---------------|
| Research Consent Form | | |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Netwo | ork Affiliates | OHRS 07.17.15 |

## B. WHY IS THIS RESEARCH STUDY BEING DONE?

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved capmatinib as a treatment for any disease.

In this research study, we are using the study drug called capmatinib. Capmatinib is a specific blocker of the cMET protein. This protein acts as a trigger to start a series of events in your cells in what is known as the C-MET pathway. By doing this, capmatinib may slow or stop the growth and/or survival of cancer cells. Capmatinib is not yet FDA approved for the treatment of people with your cancer. It is not known if capmatinib will be effective in people who have previously had other drugs that block the cMET pathway. This study will help us understand how capmatinib works in your body and what capmatinib does to your cancer. Any potential harmful effects of capmatinib will also be studied.

## C. WHAT OTHER OPTIONS ARE THERE?

Taking part in this research study is voluntary. Instead of being in this research study, you have other options which may include the following:

- Receive standard treatment including chemotherapy or immunotherapy, including FDA-approved regimens such as docetaxel and ramucirumab, or nivolumab, or pembrolizumab, which have improved overall survival in lung cancer.
- Take part in another research study.
- Receive no therapy specific to your cancer.
- Comfort care, also called palliative care. This type of care may help to reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to treat the symptoms.

Please talk to the research doctor about your options before you decide whether you will take part in this research study.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|-----------------------------------------|----------------|---------------|
| Research Consent Form | | |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Network | ork Affiliates | OHRS 07.17.15 |

## D. WHAT IS INVOLVED IN THE RESEARCH STUDY?

## Before the research starts (screening):

After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

- A medical history/physical exam, the doctor will examine you and measure your weight, and vital signs (temperature, blood pressure and heart rate)
- Collection of blood sample(s) for various safety assessments (1 teaspoon of blood will be collected). Blood sampling for research.
- An assessment of your tumor by one or more of the following standard assessment tools: CT (Computerized Tomography) scan or MRI (Magnetic Resonance Imaging)
- Archival tumor tissue will be collected if available
- Pregnancy test, blood sample
- Electrocardiogram (ECG), which measures your heartbeat

If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

In this study, a treatment cycle lasts 21 days starting from Day 1 (the first dose of study drug). You will be asked to come back to the doctor's office/clinic twice during the first cycle (first 21 days) on Day 1 and Day 8, and then every 21 days thereafter from Day 1 so that your condition can be monitored. Once you have been on the study drug for an extended period of time (up to Cycle 18 or approximately 13 months), these assessments will be performed at a decreased frequency of once every other cycle instead of once every cycle. Each visit may take a few hours depending upon the assessments and tests that need to be performed.

## The following tests and procedures will be done as long as you are enrolled in the study:

Oral Study Drug: Each treatment cycle lasts 21 days during which time you
will be taking the study drug two times per day.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm |
|-------------------------|
| Research Consent Form |
| for Diamodical Descends |

**for Biomedical Research**Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 07.17.15

- Medical history/physical examination: The doctor will examine you and measure your weight, and vital signs (temperature, blood pressure and heart rate) on Day 1 of each cycle visit and at the end of the treatment (EOT).
- Blood sampling for hematology and biochemistry: Day 1 of each cycle visit and day 8 of the first cycle. 1 teaspoon of blood will be collected for laboratory testing each time these assessments are measured.
- Blood sampling for biomarkers (ctDNA): Every two cycles and EOT.
- **Electrocardiogram (ECG)**, which measures your heartbeat on Day 1 of every cycle and EOT.
- Radiological imaging to assess your tumor: every two cycles (approximately every six weeks).
- Concomitant medications: You will be asked about any medications you have been taking. This includes prescriptions drugs, over-the-counter medicines, natural or herbal medicines, alternative medicines and vitamins.

Sometimes it is hard to keep track of all of the details and procedures that are part of a research study. We will describe them in this consent form and you can refer to this at any time during the research study.

If you take part in this research study you will be given a drug diary. You will be asked to document information in the drug diary about the study treatment you are being asked to take.

| | | | | +/- 3 day wii | ndow aroun | d visits |
|---|---|---|---|---|---|---|
| Visit Name | Screen | Cycle days ) | 1 (21 | Cycle 2-18<br>(Up to<br>Month 13) | Cycles > 18 (Months > 13) | End of<br>Treatment |
| Day of cycle | -28 to - | C1<br>D1 | C1<br>D8 | Day 1 | Day 1 of<br>Every<br>Other<br>Cycle | |
| Obtain study informed consent | x | | | | | |
| Collection of archival tumor tissue if possible | x | | | | | |
| Confirming Tissue | X | | | | | |
| Inclusion/exclusion criteria | x | | | | | |


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 0/3/2021 3.31 pm | 8/3/2021 | 9:37 | pm |
|------------------|----------|------|----|
|------------------|----------|------|----|

## Research Consent Form for Biomedical Research

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 07.17.15

| | | | | +/- 3 day window around visits | | |
|---|---|---|---|---|---|---|
| Visit Name | Screen | Cycle 1 (21 days) | | Cycle 2-18<br>(Up to<br>Month 13) | Cycles > 18 (Months > 13) | End of<br>Treatment |
| Day of cycle | -28 to - | C1<br>D1 | C1<br>D8 | Day 1 | Day 1 of<br>Every<br>Other<br>Cycle | |
| Relevant medical and oncologic history | x | | | | | |
| Physical examination | X | х | X | X | X | X |
| Vital signs | X | X | X | X | X | X |
| Performance status | X | X | X | X | X | x |
| ECG | X | X | | X | X | x |
| Pregnancy test (serum test) | X | | | | | |
| Hematology | X | X | X | X | X | X |
| Chemistry | X | X | X | X | X | x |
| Tumor evaluation<br>(CT/MRI) | X | | | Every two cy | veles | |
| Adverse events | | X | X | X | X | X |
| Optional tumor biopsy | X | | | | | X |
| Circulating tumor DNA | x | Every | two cy | cles | | x |

### Study treatment discontinuation

Please inform your doctor or study staff if you decide to interrupt or stop taking the study treatment. You will be asked to return to the study site as soon as possible and within 7 days of the last dose of capmatinib to check how you are doing and feeling. Also, the study doctor may choose to discontinue your study treatment if you are not doing well on the study drug. Upon treatment discontinuation, the following tests will be performed:

- **Physical Examination**: The doctor will examine you and measure your weight, and vital signs (temperature, blood pressure and heart rate).
- **Performance status:** your performance status will be assessed, based on how your disease affects your ability to carry out normal activities.
- Concomitant medications: You will be asked about any medications you have been taking. This includes prescriptions drugs, over-the-counter medicines, natural or herbal medicines, alternative medicines and vitamins.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|---------------------------------------|---------------|---------------|
| Research Consent Form | | |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Netwo | rk Affiliates | OHRS 07.17.15 |

- Blood sampling for hematology and biochemistry: safety assessments.
- Electrocardiogram (ECG), which measures your heartbeat.
- Radiological imaging to assess your tumor: Radiologic imaging to find and measure your tumor(s) and assess the status of your disease, if it is not done within 4 weeks prior to the day of last dose.

Regardless of the reason for discontinuation from study treatment, you will be contacted for a safety follow-up visit 30 days after the last dose of capmatinib. At this time, your doctor or study nurse will ask you how you are feeling and check on possible new symptoms or evolution of previous symptoms that have occurred after discontinuation of study treatment. You will also be asked if you have started any new anticancer therapies since discontinuing the study.

If you cannot or do not want to continue to attend study visits while off study treatment, your study doctor or study staff may ask if they can contact you by telephone until the end of the study to check on how you are doing. You may decline contact by telephone if you so choose.

### Planned Post Treatment Follow-up:

We would like to keep track of your medical condition on an annual basis. Keeping in touch with you and checking your condition every year helps us look at the long-term effects of the research study.

## E. How long will I be in this research study?

You will be in this research study for as long as there is no disease progression and/or the study doctor feels there is clinical benefit.

The research doctor may decide to take you off the research study for many reasons including if:

- It is considered to be in your best interest
- The study treatment or procedures are found to be unsafe or ineffective
- There is any problem with following study treatments and procedures
- Your condition worsens
- Or for other unforeseen reasons that make it necessary to stop your participation in the research study

If you are removed from the research study, the research doctor will explain to you why you were removed.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm |
|------------------------------------|
| Research Consent Form |
| for Biomedical Research |
| Dana-Farber/ Harvard Cancer Center |

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

In addition, you can stop participating in the research study at any time, however, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study. If you decide to stop participating in this research study, we encourage you to talk to the research doctor and your primary doctor first.

OHRS 07.17.15

## F. WHAT ARE THE RISKS OR DISCOMFORTS OF THE RESEARCH STUDY?

There are risks to taking part in any research study. One risk is that you may get a study drug that does not help treat your disease or that makes your condition or disease worse. Another risk is that there may be side effects.

All cancer treatments can have side effects, which can range from mild and reversible to severe, long lasting and possibly life-threatening. There is a great deal of variability among side effects of different cancer treatments and between individuals. In a research study, all of the risks or side effects may not be known before you start the study. You need to tell your doctor or a member of the study team immediately if you experience any side effects.

Everyone in the research study will be watched carefully for side effects. You will be monitored during the administration of study drugs to keep track of your blood counts and organ function, particularly your kidney and liver function. If you experience side effects, they may go away after you stop taking the study drug. Some side effects can be mild; but others can be long lasting and may never go away. Some may be life-threatening or fatal.

Since the effect of the study drug(s) taken with other medications may not be known, it is important that you tell the research doctor about all prescription and non-prescription drugs, herbal preparations and nutritional supplements that you are taking or planning to take. There may also be some foods that you should avoid while on this research study and your research doctor will review this information with you.

During the research study, you will be notified of newly discovered side effects or significant findings, which may affect your health or willingness to participate. You may be asked to sign a new consent form that shows that you have been informed of new information relating to this research study.

## Risks Associated with Capmatinib: Frequent: Between a 10-50% Chance


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | |
|-----------------------|---|
| Research Consent Form | · |

# for Biomedical Research Dana-Farber/ Harvard Cancer Center

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 07.17.15

- Abnormal physical weakness and/or lack of energy
- Liver enzyme (called transaminase, ALT) increase (possible sign of live dysfunction)
- Chest pain
- Decreased appetite
- Diarrhea
- Nausea
- Vomiting
- Fatigue
- Swelling in arms and legs (Peripheral edema)
- Blood creatinine increase (a measure of how well your kidney is working)
- Constipation
- Low levels of a blood protein called albumin, which can cause generalized swelling, edema (Hypoalbuminemia)
- Fever
- Low number of red blood cells that can cause tiredness and shortness of breath- may require a blood transfusion (Anemia)
- Cough
- Difficulty breathing
- Abnormal digestive blood test (Lipase increase- no symptoms or sweating/weakness/pain/nausea/vomiting if pancreas function is affected)
- Abnormal blood test- possible pancreas damage (Amylase increasewhich may manifest as symptoms such as nausea, vomiting or pain)
- Back, joint, muscle, ligament, tendon, and bone pain (Musculoskeletal pain)

#### Occasional: Between a 5-10% chance

- Bacterial skin infection with redness of the skin (cellulitis)
- Abnormal liver test- possible liver damage (AST and/or gammaglutamyltransferase (GGT) increase- which may manifest as symptoms such as fatigue, nausea, abdominal pain)
- Build up of fluid in the abdomen, which causes bloating and discomfortthis could require that the fluid be removed by a procedure called paracentesis (Ascites)
- Abdominal distension (another form of abdominal swelling)
- Insomnia

#### 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm |
|-------------------------|
| Research Consent Form |
| for Biomedical Research |

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 07.17.15

- Blood bilirubin increase (substance that is usually removed from body by feces- symptom can be yellowing of the skin and whites of the eyes (Jaundice)
- Decreased levels of sodium in the blood, which can cause confusion, seizures, fatigue and low levels of consciousness (Hyponatraemia)
- Severe skin itch
- Tremor
- Indigestion
- Interstitial lung disease (a type of inflammation of lung tissue also called ILD or pneumonitis) which can cause shortness of breath and difficulty breathing. If severe, this can be life threatening. It is important that you alert your doctor of any signs of breathing difficulties or new onset of cough while taking the study medication.
- Impairment of kidney function (renal impairment)
- Skin rash with red, raised itchy bumps/hives (urticaria)

### **Uncommon (less than 5% chance):**

- Dizziness
- Acute renal failure (kidney failure which is when both of your kidneys fail
  and your body holds fluid which can be serious or life threatening- your
  blood pressure rises and harmful wastes build up in your body- you may
  experience fatigue, nausea, and loss of appetite- when this happens, you
  need treatment to replace the work of your failed kidneys such as dialysis)
- This study treatment may cause low blood cell counts (white blood cells).
- Sudden painful, inflammation of the pancreas (acute pancreatitis)
- Headache
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and/or difficulty breathing. (Neutropenia)
- Elevation of alkaline phosphatase, an enzyme of liver and bone, might indicate damage to liver or bone. You may experience no symptoms related to this abnormal laboratory finding.

Cancer research often includes scans and x-rays that are also provided as routine care. The following describes the side effects of procedures done only for the purposes of research.

#### 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm |
|--------------------------------------------------|
| Research Consent Form<br>for Biomedical Research |

OHRS 07.17.15

## Radiation Risks Associated with Scans and X-Rays:

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

While you are in this research study, CT scans may be used to evaluate your disease. The frequency of these exams is slightly greater than what you would receive as standard care. In the long term, over many years, there is a very low risk of developing a new cancer as a result of the radiological evaluation and treatment for your cancer. Certain types of drugs or combinations of these drugs with radiation may further slightly increase the risk of developing a new cancer.

### Risks Associated with MRI Scans:

Dana-Farber/ Harvard Cancer Center

When having an MRI (Magnetic Resonance Imaging) scan, you will lie still on a table that slides into a tunnel slightly wider than your body. People who feel uncomfortable in confined spaces (claustrophobia) may feel uncomfortable in the narrow cylinder. If you feel uncomfortable in confined spaces, please tell your research doctor. Your doctor may give you a medication to make you feel more comfortable. As images are taken, a loud banging noise will be produced. Earplugs or headphones will be available if needed. The MRI can be stopped at any time at your request, but the scan may not be complete.

### Risks Associated with Contrast Agents Used During Scans:

There is a small risk with using a contrast agent that is injected into a vein during the CT scan and MRI. The contrast agent is a special dye that highlights organs, blood vessels or tissue to make them more visible. Depending on the type of contrast agent that is used, it may cause decreased kidney function or worsen kidney function in people who already have decreased kidney function. Therefore, we will monitor your kidney function closely while you participate in this study. If there is any change in your kidney function, we may have to remove you from the study.

Uncommonly, some people have allergic reactions (such as hives and itching) to the contrast agent. Serious reactions (for example, drop in blood pressure, difficulty breathing or severe allergic reaction and death) are rare.

### **Reproductive Risks:**

The drugs used in this research study may affect a fetus. While participating in this research study, you should not become pregnant or father a baby, and should not nurse a baby. We can provide counseling about preventing pregnancy for either male or female study participants. Let your doctor know immediately if you become pregnant or find out that you are going to be the father of a child.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm |
|------------------------------------|
| Research Consent Form |
| for Biomedical Research |
| Dana-Farber/ Harvard Cancer Center |

#### Non-Physical Risks:

Because of side effects or the time required for tests and clinic visits while you are on this research study, you may be unable to keep up with your normal daily activities.

OHRS 07.17.15

## G. WHAT ARE THE BENEFITS OF THE RESEARCH STUDY?

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

This study may or may not help you. This study may help researchers learn things that may help people in the future.

## H. CAN I STOP BEING IN THE RESEARCH STUDY AND WHAT ARE MY RIGHTS?

You have the right to choose not to sign this form. If you decide not to sign this form, you cannot participate in this research study.

You can stop being in the research study at any time. Tell the research doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop. Leaving the research study will not affect your medical care outside of the research study.

If you choose not to participate, are not eligible to participate, or withdraw from this research study, this will not affect your present or future care and will not cause any penalty or loss of benefits to which you are otherwise entitled.

It is important to tell the research doctor if you are thinking about stopping so your research doctor can evaluate the risks from stopping the capmatinib drug. In some cases, the abrupt stopping of a drug can have risks in itself. Another reason to tell your research doctor that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

## I. WILL I BE PAID TO TAKE PART IN THIS RESEARCH STUDY?

You will not receive payment for participating in this study.

## J. WHAT ARE THE COSTS?

Taking part in this research study might lead to added costs to you or your insurance company.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |



Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 07.17.15

You will not be charged for capmatinib.

You or your insurance company will be charged for portions of your care during this research study that are considered standard care. You may be responsible for co-payments and deductibles that are typical for your insurance coverage.

If you have questions about your insurance coverage, or the items you might be required to pay for, please call financial services for information. The contact information for financial services are:

- Beth Israel Deaconess Medical Center: (617) 667-5661
- Massachusetts General Hospital: (617) 726-2191

The National Cancer Institute provides an online resource to help people participating in cancer clinical trials understand which services their insurance company is required by law to pay. This can be found at the website below or can be provided by the study team:

www.cancer.gov or 1-800-4-CANCER (1-800-422-6237)

## K. WHAT HAPPENS IF I AM INJURED OR SICK BECAUSE I TOOK PART IN THIS RESEARCH STUDY?

If you think you have been injured as a result of taking part in this research study, tell the person in charge of this research study as soon as possible. The research doctor's name and phone number are listed in this consent form.

The treating hospital will offer you the care needed to treat injuries directly resulting from taking part in this research. The treating hospital may bill your insurance company or other third parties, if appropriate, for the costs of the care you get for the injury, but you may also be responsible for some of them.

There are no plans for any of the sponsors of this study or Novartis to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

We will need to collect certain personal information about you for insurance or payment reporting purposes, such as your name, date of birth, gender, social security number or Medicare identification number and information related to this


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |



OHRS 07.17.15

research study. We may be required to report this information to the Centers for Medicare & Medicaid Services. We will not use this information for any other purpose.

## L. WHAT ABOUT CONFIDENTIALITY?

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

Dana-Farber/ Harvard Cancer Center

We will take measures to protect the privacy and security of all your personal information, but we cannot guarantee complete confidentiality of study data.

Medical information created by this research study may become part of your hospital medical record and may be forwarded to your primary doctor. Information that does not become part of your medical record will be stored in your study file.

The results of this research study may be published. You will not be identified in publications without your permission.

The drug supplier of this research study, Novartis Pharmaceuticals may use health information about you to do the research described in this form and for related research. However, this information does not include your name. Related research means research related to the drug capmatinib and/or the medical condition studied here, cancer, which is the same disease area being studied in this research.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## M. FINANCIAL DISCLOSURES

It is possible that certain researchers on this study may have earned money from, or own some publicly-traded stock in, the company that makes or is developing the study drug capmatinib. The amount of money that a researcher may earn and still take part in research is limited by the Harvard Medical School Faculty of Medicine Policy on Conflicts of Interest and Commitment. If you have further questions, please speak with a member of the study team or contact the Dana-Farber Cancer Institute Office of Research Integrity at 617-432-4557 or researchintegrity@dfci.harvard.edu.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|--------------------------------------|----------------|---------------|
| Research Consent Form | | |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Netw | ork Affiliates | OHRS 07.17.15 |

## N. WHOM DO I CONTACT IF I HAVE QUESTIONS ABOUT THE RESEARCH STUDY?

If you have questions about the study, please contact the research doctor or study staff as listed below:

Massachusetts General Hospital

• Rebecca S. Heist, MD: 617-724-4000

Beth Israel Deaconess Medical Center

Daniel Botelho Costa, MD, PhD, MMSc: 617-667-9236

24-hour contact for questions about the study or to report a study-related injury after hospital hours, please call Massachusetts General Hospital at 617-724-4000 and ask your doctor to be paged.

For questions about your rights as a research participant, please contact a representative of the Office for Human Research Studies at DFCI (617) 632-3029. This can include questions about your participation in the study, concerns about the study, a research related injury, or if you feel/felt under pressure to enroll in this research study or to continue to participate in this research study.

## O. PRIVACY OF PROTECTED HEALTH INFORMATION

Federal law requires Dana-Farber/Harvard Cancer Center (DF/HCC) and its affiliated research doctors, health care providers, and physician network to protect the privacy of information that identifies you and relates to your past, present, and future physical and mental health conditions ("protected health information"). If you enroll in this research study, your "protected health information" will be used and shared with others as explained below.

## 1. What protected health information about me will be used or shared with others during this research?

- Existing medical records, including mental health records.
- New health information created from study-related tests, procedures, visits, and/or questionnaires

#### 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|--------------------------------------|----------------|---------------|
| Research Consent Form | | Ī |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Netw | ork Affiliates | OHRS 07.17.15 |

## 2. Why will protected information about me be used or shared with others?

The main reasons include the following:

- To conduct and oversee the research described earlier in this form;
- To ensure the research meets legal, institutional, and accreditation requirements;
- To conduct public health activities (including reporting of adverse events or situations where you or others may be at pne of harm); and
- To provide the study sponsor and the drug supplier with information arising from an adverse event or other event that relates to the safety or toxicity of the drug for the purpose of this or other research relating the study drug and its use in cancer; and,
- Other reasons may include for treatment, payment, or health care operations. For example, some medical information produced by this research study may become part of your hospital medical record because the information may be necessary for your medical care. (You will also be given a notice for use and sharing of protected health information.)

### 3. Who will use or share protected health information about me?

 DF/HCC and its affiliated research doctors and entities participating in the research will use and share your protected health information. In addition, other DF/HCC offices that deal with research oversight, billing or quality assurance will be able to use and share your protected health information.

## 4. With whom outside of DF/HCC may my protected health information be shared?

While all reasonable efforts will be made to protect the confidentiality of your protected health information, it may also be shared with the following entities:

- Outside individuals or entities that have a need to access this information to perform functions relating to the conduct of this research such as analysis by outside laboratories on behalf of DF/HCC and its affiliates (for example, data storage companies, insurers, or legal advisors).
- The drug supplier of the study, its subcontractors and its agent(s):
   Novartis and its authorized agents
- Other research doctors and medical centers participating in this research, if applicable


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm |
|-------------------------|
| Research Consent Form |
| for Biomedical Research |

OHRS 07.17.15

- Federal and state agencies (for example, the Department of Health and Human Services, the Food and Drug Administration, the National Institutes of Health, and/or the Office for Human Research Protections), or other domestic or foreign government bodies if required by law and/or necessary for oversight purposes. A qualified representative of the FDA and the National Cancer Institute may review your medical records.
- Hospital accrediting agencies

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

Dana-Farber/ Harvard Cancer Center

 A data safety monitoring board organized to oversee this research, if applicable

Some who may receive your protected health information may not have to satisfy the privacy rules and requirements. They, in fact, may share your information with others without your permission.

## 5. For how long will protected health information about me be used or shared with others?

 There is no scheduled date at which your protected health information that is being used or shared for this research will be destroyed, because research is an ongoing process.

## 6. Statement of privacy rights:

- You have the right to withdraw your permission for the research doctors and participating DF/HCC entities to use or share your protected health information. We will not be able to withdraw all the information that already has been used or shared with others to carry out related activities such as oversight, or that is needed to ensure quality of the study. To withdraw your permission, you must do so in writing by contacting the researcher listed above in the section: "Whom do I contact if I have questions about the research study?"
- You have the right to request access to your protected health information that is used or shared during this research and that is related to your treatment or payment for your treatment, but you may access this information only after the study is completed. To request this information, please contact the researcher listed above in the section: "Whom do I contact if I have questions about the research study?"

#### 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|--------------------------------------|-----------------|---------------|
| Research Consent Form | | |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer Center | | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Netw | vork Affiliates | OHRS 07.17.15 |

## P. OPTIONAL RESEARCH STUDY:

You are being asked to participate in some optional research. If you decide not to participate in the optional research, you can still participate in the main research study. Please take your time to make your decision and discuss it with others and your primary care physician. Your participation in this optional research is voluntary, and you will not be penalized or lose any benefits if you refuse to participate or decide to stop.

### Optional Study:

A biopsy will be collected pre-dose during screening and at End of Treatment (EOT). These biopsies will be assessed by techniques such as Next Generation Sequencing (NGS) to assess potential mechanisms of sensitivity and resistance to capmatinib therapy. NGS performs DNA sequencing, during which millions of fragments of DNA from a single sample are sequenced together at once. These results are exploratory only and will not be available in real time. However results that may be applicable to you will be shared with your treating physician who will share them with you. Only those results which are performed in a CLIA certified laboratory will be shared, all other studies are exploratory research only.

## Risks Associated with Biopsies:

Biopsies are normally performed under the guidance of an imaging technique. Each procedure requires a separate consent prior to the biopsy. The risks may include:

- Pain and discomfort. The amount of pain and discomfort will vary, depending on the location of the biopsy site. These risks can be discussed with the study doctor.
- Minor bleeding at the biopsy site.
- Tenderness at the biopsy site.
- Scarring at the biopsy site.
- Rarely, an infection at the biopsy site.

Uncommonly, complications from biopsies can be life threatening. As with any interventional procedure, other potentially serious complications from bleeding or organ damage may occur. These might require additional surgical intervention.

You will not be charged for this optional study.


| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|---|---|---|
| Research Consent Form<br>for Biomedical Research<br>Dana-Farber/ Harvard Cancer Cer | | |
| BIDMC/BCH/BWH/DFCI/MGH/ | Partners Network Affiliates | OHRS 07.17.15 |
| Please indicate whether of screening and EOT (End | or not you want to take part in the of Treatment). | optional biopsies at |
| □ Yes | Initials | Date |
| □ No | Initials | Date |

## 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:37 pm | | |
|---|---|---|
| Research Consent Form for Biomedical Research Dana-Farber/ Harvard Cancer Center | 1 4 651. | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Netv | WOLK ATTITIATES | OHRS 07.17.15 |
| Q. DOCUMENTATION OF CONSENT | | |

My signature below indicates:

- I have had enough time to read the consent and think about participating in this study;
- I have had all of my questions answered to my satisfaction;
- I am willing to participate in this study;
- I have been told that my participation is voluntary and I can withdraw at any time

| Signature of Participant or Legally Authorized Representative | Date |
|---|---|
| Relationship of Legally Authorized Repres | sentative to Participant |

## 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |

| 8/3/2021 9:3 | <i>i</i> / | pm |
|--------------|------------|----|
|--------------|------------|----|

## **Research Consent Form for Biomedical Research**

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 07.17.15

| Adult Participants |
|---|
| To be completed by person obtaining consent: |
| The consent discussion was initiated on (date). |
| Signature of individual obtaining consent: |
| Printed name of above: |
| Date: A copy of this signed consent form will be given to the participant or legally authorized representative, or, where the participant is a minor, the participant's parent or legal guardian. |
| For Adult Participants |
| 1) The participant is an adult and provided consent to participate. |
| 1a) Participant (or legally authorized representative) is a non-English speaker and signed the translated Short Form in lieu of English consent document: |
| As someone who understands both English and the language spoken by the participant, I interpreted and/or witnessed, in the participant's language, the researcher's presentation of the English consent form. The participant was given the opportunity to ask questions. |
| Signature of Interpreter/Witness: |
| Printed Name of Interpreter/Witness: |
| Date: 1b) Participant is illiterate |
| The consent form was read to the participant who was given the opportunity to ask questions. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: |
| <ul> <li>2) The participant is an adult who lacks capacity to provide consent and his/her legally<br/>authorized representative:</li> </ul> |
| <ul><li>2a) gave permission for the adult participant to participate</li></ul> |
| <ul><li>2b) did not give permission for the adult participant to participate</li></ul> |

## 

| DFCI Protocol Number: | 16-019 | Approved Date (DFCI IRB Approval): | 02/06/2020 |
|---|---|---|---|
| Date Posted for Use: | 02/11/2020 | | |